CLINICAL TRIAL: NCT02309112
Title: Yoga for Health-related Quality of Life in Adult Cancer: A Randomized Controlled Feasibility Trial
Brief Title: Yoga in Adult Cancer: A Feasibility Trial
Acronym: Y-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of British Columbia (Other); British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OXTREC 534-14
Record Dates: First submitted 2014-11-21; First posted 2014-12-05 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2014-11

CONDITIONS: Quality of Life
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Yoga Group A: Minimum Exposure (Experimental): The minimum-exposure yoga package, this intervention included 45-minutes of contact time with a trained yoga professional. In Week 1, this session included a 30-minute introductory session focussing on pranayama (breathing techniques), as well as a brief introduction to available community-based and online yoga to encourage a safe home-based practice (15-minutes). Financial subsidy, compensation or special promotion of any particular yoga was not provided. Participants were invited to stay for a social discussion following the yoga class.
  Interventions: Other: Yoga
- Yoga Group B: Medium Exposure (Experimental): The medium-exposure yoga package, this intervention included the components of Group A, with an additional 30-minute orientation and safety training of how to practice yoga dhyana (meditation techniques) and asana (physical postures) in Week 1. Participants were then invited to stay and ask questions following the yoga class. A pre-paid online yoga membership to http://www.myyogaonline.com was offered for the duration of the study (Weeks 1 to 4). In addition to this, one 120-minute workshop to further develop yoga pranayama, dhyana and asana training was administered by an expert instructor during Week 2 or 3.
  Interventions: Other: Yoga
- Yoga Group C: Maximum Exposure (Experimental): The maximum-dose yoga package, this intervention includes the components of Group A, with the same 30-minute orientation and safety training of how to practice yoga dhyana (meditation techniques) and asana (physical postures) in Week 1. Participants were invited to stay and ask questions following the yoga class. As in Group B, a pre-paid online yoga membership to http://www.myyogaonline.com was also provided for the duration of the study (Weeks 1 to 4). Participants were then invited to attend three 60-minute yoga group classes led by an expert yoga instructor per week (Weeks 1 to 4). These yoga sessions were held in a clinical setting in proximity to their treatment location and delivered at no cost to the patient.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — A mind-body therapy that includes specified breathing, meditation and physical postures.

SUMMARY:
A feasibility study to determine the appropriateness of yoga intervention to improve health-related quality of life in adult cancer patients.

DETAILED DESCRIPTION:
A prospective, mixed methods feasibility trial allocated participants to receive one of three yoga interventions over a four-week study period. Data collection was completed through online survey of QOL-CA/CS and customized surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult cancer patients 19 years of age or older
2. Patients receiving or planning to receive conventional treatment that includes at least one of chemotherapy, radiotherapy, hormone therapy or active surveillance within 28 days
3. Patients in any stage of cancer diagnoses of all tumour types and locations
4. Participants with internet access and willingness to participate in online communication
5. Participants with access to transportation and personal willingness to attend meetings in central Vancouver, Canada.
6. Participants fluent in the English language

Exclusion Criteria:

1. Patients with any physical limitation, risk of personal injury or under proscription of light to moderate physical activity
2. Patients with pre or post surgical interventions were excluded due to potential physical limitations or safety concerns with wound healing
3. Regular or experienced practitioners of yoga were excluded and defined as those patients reporting current or historical use of regular yoga (>2 session per month in past 12 months)
4. Patients undergoing medical treatment for serious psychological disturbances that might have interfered with adherence to protocol and/or ability to provide informed consent were excluded (e.g. multiple personality disorders, severe depression, obsessive-compulsive disorder)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie McDonald, MSW, Principal Investigator — Vancouver-BCCA

REFERENCES:
- [Derived] McCall M, McDonald M, Thorne S, Ward A, Heneghan C. Yoga for Health-Related Quality of Life in Adult Cancer: A Randomized Controlled Feasibility Study. Evid Based Complement Alternat Med. 2015;2015:816820. doi: 10.1155/2015/816820. Epub 2015 Jun 11. PMID 26170884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in Vancouver, Canada commenced on April 15, 2014 via poster advertisements in Vancouver cancer clinics (n=3).
Pre-assignment Details: No wash out or run-in period was allocated.
  Recruitment ended on June 30, 2014 and participants were randomized on July 1, 2014.
Groups:
- Yoga Group A: The minimum-exposure yoga package, this intervention included 45-minutes of contact time with a trained yoga professional. This session included a 30-minute introductory session focussing on pranayama (breathing techniques), as well as a brief introduction to available community-based and online yoga to encourage a safe home-based practice (15-minutes). Financial subsidy, compensation or special promotion of any particular yoga was not provided. Participants were invited to stay for a social discussion following the yoga class.
  Yoga: A mind-body therapy that includes specified breathing, meditation and physical postures.
- Yoga Group B: The medium-exposure yoga package, this intervention includes the components of Group A, with an additional 30-minute orientation and safety training of how to practice yoga dhyana (meditation techniques) and asana (physical postures) in week one. Participants were invited to stay and ask questions following the yoga class. A pre-paid online yoga membership to http://www.myyogaonline.com was offered for the duration of the study. In addition to this, one 120-minute workshop to further develop yoga pranayama, dhyana and asana training was administered by an expert instructor during week 2 or 3.
  Yoga: A mind-body therapy that includes specified breathing, meditation and physical postures.
- Yoga Group C: The maximum-dose yoga package, this intervention includes the components of Group A, with the same 30-minute orientation and safety training of how to practice yoga dhyana (meditation techniques) and asana (physical postures) in week one. Participants were invited to stay and ask questions following the yoga class. As in Group B, a pre-paid online yoga membership to http://www.myyogaonline.com was also provided for the duration of the study. Participants were then invited to attend three 60-minute yoga group classes led by an expert yoga instructor per week (weeks 1 to 4). These yoga sessions were held in a clinical setting in proximity to their treatment location and delivered at no cost to the patient.
  Yoga: A mind-body therapy that includes specified breathing, meditation and physical postures.
Period: Overall Study
Arm/Group | Yoga Group A | Yoga Group B | Yoga Group C
Started | 5 | 5 | 5
Completed Yoga Intervention | 4 | 5 | 4
Completed | 4 | 4 | 4
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The sample includes male and female (n=11) adult cancer patients receiving conventional treatment in Vancouver, Canada.
  Patients undergoing one or more treatments of chemotherapy, radiation, hormone therapy or active surveillance were included in the study. Baseline data collection included all types of treatment for a primary cancer diagnosis.
Groups:
- Yoga Group A: Minimum Exposure: The minimum-exposure yoga package, this intervention included 45-minutes of contact time with a trained yoga professional. This session included a 30-minute introductory session focussing on pranayama (breathing techniques), as well as a brief introduction to available community-based and online yoga to encourage a safe home-based practice (15-minutes). Financial subsidy, compensation or special promotion of any particular yoga was not provided. Participants were invited to stay for a social discussion following the yoga class.
  Yoga: A mind-body therapy that includes specified breathing, meditation and physical postures.
- Yoga Group B: Medium Exposure: The medium-exposure yoga package, this intervention includes the components of Group A, with an additional 30-minute orientation and safety training of how to practice yoga dhyana (meditation techniques) and asana (physical postures) in week one. Participants were invited to stay and ask questions following the yoga class. A pre-paid online yoga membership to http://www.myyogaonline.com was offered for the duration of the study. In addition to this, one 120-minute workshop to further develop yoga pranayama, dhyana and asana training was administered by an expert instructor during week 2 or 3.
  Yoga: A mind-body therapy that includes specified breathing, meditation and physical postures.
- Yoga Group C: Maximum Exposure: The maximum-dose yoga package, this intervention includes the components of Group A, with the same 30-minute orientation and safety training of how to practice yoga dhyana (meditation techniques) and asana (physical postures) in week one. Participants were invited to stay and ask questions following the yoga class. As in Group B, a pre-paid online yoga membership to http://www.myyogaonline.com was also provided for the duration of the study. Participants were then invited to attend three 60-minute yoga group classes led by an expert yoga instructor per week (weeks 1 to 4). These yoga sessions were held in a clinical setting in proximity to their treatment location and delivered at no cost to the patient.
  Yoga: A mind-body therapy that includes specified breathing, meditation and physical postures.
- Total: Total of all reporting groups
Arm/Group | Yoga Group A: Minimum Exposure | Yoga Group B: Medium Exposure | Yoga Group C: Maximum Exposure | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Full Range); unit: years] | 51.6 [41 to 66] | 57.2 [43 to 72] | 45 [33 to 57] | 51.3 [33 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 5 | 5 | 15
Tumour Location [Number; unit: participants]
  Breast | 3 | 1 | 2 | 6
  Prostate | 0 | 1 | 1 | 2
  Colorectal | 1 | 1 | 0 | 2
  Blood | 0 | 0 | 1 | 1
  Skin | 0 | 1 | 0 | 1
  Abdomen | 0 | 1 | 0 | 1
  Tongue | 1 | 0 | 0 | 1
  Brain | 0 | 0 | 1 | 1
Stage of Cancer Diagnosis [Number; unit: participants]
  Stage I | 2 | 1 | 1 | 4
  Stage II | 2 | 0 | 1 | 3
  Stage III | 1 | 2 | 2 | 5
  Stage IV | 0 | 1 | 0 | 1
  not reported | 0 | 1 | 1 | 2
Types of Conventional Treatment [Number; unit: participants] — Participants were asked to self-report any and all aspects of current conventional treatments for their cancer diagnosis; multiple treatments were recorded (i.e. radiotherapy, chemotherapy, hormone therapy or active surveillance)
  participants
    Chemotherapy | 3 | 2 | 2 | 7
    Radiotherapy | 3 | 3 | 2 | 8
    Hormone Therapy | 2 | 2 | 1 | 5
    Active Surveillance | 1 | 2 | 2 | 5
    Post-surgical Intervention | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Patient Recruitment to Yoga Intervention
Description: Number of participants eligible for randomization to yoga intervention during cancer treatment
Time Frame: 10 weeks
Population: Male (n=4) and female (n=11) adult patients undergoing conventional treatment in Vancouver, Canada for a cancer diagnosis; who have not participated in yoga the past month.
Measure: Number; unit: participants
Groups:
- Eligible Participants: The group of eligible participants who agreed to be randomized to ono of three yoga groups.
Arm/Group | Eligible Participants
Number analyzed (Participants) | 15
participants
  Number of participants randomized to yoga | 15
  Rate of patient recruitment per week | 1.5

2. Secondary Outcome: Patient Adherence to Yoga Intervention
Description: Number of participants who completed their yoga intervention
Time Frame: 6 weeks
Population: Male (n=4) and female (n=11) adult patients undergoing conventional treatment for cancer diagnosis in Vancouver, Canada
Measure: Number; unit: participants
Groups:
- Yoga Group A: Minimum Exposure: Week 1: 1 x 45-minute introductory yoga session (breathing techniques only); recommended community-based resources for in-person yoga and online yoga; equipment to encourage a home-based practice (i.e illustrated manual, yoga mat)
- Yoga Group B: Medium Exposure: Week 1: 1 x 75-minute introductory yoga session (breathing, meditation and physical postures); recommended community-based resources for in-person yoga; equipment to encourage a home-based practice (i.e illustrated manual, yoga mat) Weeks 1 to 4: pre-paid online yoga Week 2 or 3: 1 x 120-minute yoga session (breathing, meditation and physical postures)
- Yoga Group C: Maximum Exposure: Week 1: 1 x 75-minute introductory yoga session (breathing, meditation and physical postures); recommended community-based resources for in-person yoga and; equipment to encourage a home-based practice (i.e illustrated manual, yoga mat) Weeks 1 to 4: pre-paid online yoga; 3 x 60-minute yoga sessions (breathing, meditation and physical postures)
Arm/Group | Yoga Group A: Minimum Exposure | Yoga Group B: Medium Exposure | Yoga Group C: Maximum Exposure
Number analyzed (Participants) | 5 | 5 | 5
participants | 4 | 5 | 4

3. Other Pre Specified Outcome: Patient Acceptability of Yoga Intervention
Description: Amount of satisfaction for adult cancer patients assessed via Likert-scale surveys; on scale of 1 to 10, 1 being not satisfied; 10 being extremely satisfied (i.e higher number, better outcome).
Time Frame: 6 weeks
Population: Adult male (n=3) and female (n=9) cancer patients undergoing conventional treatment for cancer diagnosis in Vancouver, Canada
Measure: Mean (Full Range); unit: units on satisfaction scale
Arm/Group | Yoga Group A: Minimum Exposure | Yoga Group B: Medium Exposure | Yoga Group C: Maximum Exposure
Number analyzed (Participants) | 4 | 4 | 4
units on satisfaction scale | 6.8 [1 to 10] | 7 [5 to 8] | 8.5 [6 to 10]

4. Other Pre Specified Outcome: Financial Cost of Delivering Yoga Intervention in a Clinical Setting
Description: Calculation of the per participant cost of three types of yoga interventions (Group A, B and C). The financial data included cost of in-person instruction, cost of materials and time to design and implement intervention per participant in each yoga group.
Time Frame: 10 weeks
Population: Male (n=3) and female (n=10) adult patients undergoing conventional treatment for cancer diagnosis in Vancouver, Canada
Measure: Number; unit: dollars (USD)
Groups:
- Yoga Group C: Maximum Exposure: Maximum Yoga Dose
  Week 1: 1 x 75-minute introductory yoga session (breathing, meditation and physical postures); recommended community-based resources for in-person yoga and; equipment to encourage a home-based practice (i.e illustrated manual, yoga mat) Weeks 1 to 4: pre-paid online yoga; 3 x 60-minute yoga sessions (breathing, meditation and physical postures)
Arm/Group | Yoga Group A: Minimum Exposure | Yoga Group B: Medium Exposure | Yoga Group C: Maximum Exposure
Number analyzed (Participants) | 4 | 5 | 4
dollars (USD) | 196 | 243 | 360

5. Other Pre Specified Outcome: Patient's Health-related Quality of Life
Description: Assessed via an online survey of a validated, cancer-specific survey instrument measuring health-related quality of life (QOL-CA/CS), (0 worst; 10 best possible). The QOL-CA/CS score was assessed pre and post yoga intervention.
Time Frame: 6 weeks
Population: Male (n=3) and female (n=9) adults undergoing conventional treatment for cancer diagnosis in Vancouver, Canada.
Measure: Mean (Full Range); unit: units on quality of life scale
Arm/Group | Yoga Group A: Minimum Exposure | Yoga Group B: Medium Exposure | Yoga Group C: Maximum Exposure
Number analyzed (Participants) | 4 | 4 | 4
units on quality of life scale
  Pre-intervention QOL-CA/CS | 4.88 [3.51 to 6.05] | 6.13 [5.13 to 7.9] | 5.37 [3.78 to 6.88]
  Post-intervention QOL-CA/CS | 5.54 [2.76 to 8.00] | 6.06 [4.73 to 7.25] | 5.53 [3.78 to 7.13]
  Mean Difference | 0.66 [-0.75 to 2.24] | -0.07 [-0.65 to 1.08] | 0.64 [-0.24 to 0.85]

6. Secondary Outcome: Patient Adherence Rate to Yoga Intervention
Description: % of patients who completed their yoga intervention
Time Frame: 6 weeks
Population: Male (n=4) and female (n=11) adult patients undergoing conventional treatment for cancer diagnosis in Vancouver, Canada
Measure: Number; unit: percentage of participants
Arm/Group | Yoga Group A: Minimum Exposure | Yoga Group B: Medium Exposure | Yoga Group C: Maximum Exposure
Number analyzed (Participants) | 5 | 5 | 5
percentage of participants | 80 | 100 | 80

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Self-reported injury or pain related to the yoga intervention
Arm/Group | Yoga Group A | Yoga Group B | Yoga Group C
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
As a feasibility study, the sample size is underpowered and quantitative results are unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No